CLINICAL TRIAL: NCT02261064
Title: Influence of Food on the Bioavailability of Telmisartan 40 mg/Amlodipine 5 mg Fixed-dose Combination and of Telmisartan 80 mg/Amlodipine 5 mg Fixed-dose Combination in Healthy Japanese Male Volunteers (a Phase I, Open-label, Randomised, Single-dose, Two-way Crossover Trial)
Brief Title: Influence of Food on the Bioavailability of Telmisartan/Amlodipine Fixed Dose Combination in Healthy Japanese Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1235.27
Record Dates: First submitted 2014-10-09; First posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; Amlodipine

ARMS (4):
- Telmisartan/Amlodipine low dose, fed (Experimental): Telmisartan low dose/Amlodipine fixed-dose combination
  Interventions: Drug: Telmisartan/Amlodipine low dose; Other: Japanese meal
- Telmisartan/Amlodipine low dose, fasted (Active Comparator): Telmisartan low dose/Amlodipine fixed-dose combination
  Interventions: Drug: Telmisartan/Amlodipine low dose
- Telmisartan/Amlodipine high dose, fed (Experimental): Telmisartan high dose/Amlodipine fixed-dose combination
  Interventions: Drug: Telmisartan/Amlodipine high dose; Other: Japanese meal
- Telmisartan/Amlodipine high dose, fasted (Active Comparator): Telmisartan high dose/Amlodipine fixed-dose combination
  Interventions: Drug: Telmisartan/Amlodipine high dose

INTERVENTIONS:
Drug: Telmisartan/Amlodipine low dose
  Arms: Telmisartan/Amlodipine low dose, fasted; Telmisartan/Amlodipine low dose, fed
Drug: Telmisartan/Amlodipine high dose
  Arms: Telmisartan/Amlodipine high dose, fasted; Telmisartan/Amlodipine high dose, fed
Other: Japanese meal
  Arms: Telmisartan/Amlodipine high dose, fed; Telmisartan/Amlodipine low dose, fed

SUMMARY:
Study to investigate the relative bioavailability and pharmacokinetics of the fixed-dose combination tablets (telmisartan 40 mg/amlodipine 5 mg and telmisartan 80 mg/amlodipine 5 mg) in the fed condition compared with those of the same fixed-dose combination in the fasting condition in healthy Japanese male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers without any clinically significant findings and complications on the basis of a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate, body temperature), 12-lead electrocardiograms (ECGs), clinical laboratory tests
2. Age: ≥20 and Age ≤35 years
3. Body weight: ≥50 kg
4. Body mass index (BMI): ≥18.0 and ≤25.0 kg/m2
5. Signed and dated written informed consent prior to admission to the trial in accordance with the Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
2. Diseases of the central nervous system (such as epilepsy) or psychiatric or neurological disorders
3. Chronic or relevant acute infections
4. Any clinical relevant findings in laboratory test results deviating from normal
5. A positive result in hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, a syphilitic test, or an human immunodeficiency virus (HIV) test
6. History of surgery of the gastrointestinal tract (except appendectomy)
7. History of relevant orthostatic hypotension, fainting spells, or blackouts
8. Known hypersensitivity to any component of the formulation (telmisartan and amlodipine), to any other angiotensin II receptor blockers, or to any other dihydropyridine compound
9. Intake of drugs with a long half-life (≥24 hours) within at least 1 month or less than 10 half-lives of the respective drug before drug administration
10. Intake of drugs which might reasonably influence the results of the trial on the basis of the knowledge at the time of protocol preparation within 7 days before drug administration
11. Participation in another trial with an investigational drug within 4 months or 6 half-lives of the investigational products before drug administration
12. Smoker (≥20 cigarettes/day)
13. Alcohol abuse (60 g or more ethanol/day: e.g., 3 middle-sized bottles of beer, 3 gous [equivalent to 540 mL] of sake)
14. Drug abuse
15. Blood donation (more than 100 mL within 4 weeks before drug administration)
16. Excessive physical activities (within 1 week before drug administration)
17. Intake of alcohol within 2 days before drug administration
18. Inability to comply with dietary regimen of the study centre
19. Inability to refrain from smoking during trial days
20. Subjects judged to be inappropriate by the investigator or a sub-investigator

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-12; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz) | up to 144 hours after drug administration
Maximum measured concentration of the analyte in plasma (Cmax) | up to 144 hours after drug administration

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 144 hours after drug administration
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | up to 144 hours after drug administration
Terminal rate constant of the analyte in plasma (λz) | up to 144 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | up to 144 hours after drug administration
Mean residence time of the analyte in the body after po administration (MRTpo) | up to 144 hours after drug administration
Number of subjects with adverse events | up to 56 days